CLINICAL TRIAL: NCT04855461
Title: Understanding the Determinants of Physical Activity Levels in Persons With Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Other Study IDs: EC1_CWT
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Chronic Pain
Keywords: Physical Activity; Fear of Movement; Patterns of activity; Psychological status
MeSH Terms: conditions — Chronic Pain; Motor Activity; Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed research topic will investigate the determinants of physical activity (PA) levels in patients with chronic pain. The aim of the research project is to quantify the self-reported and free-living physical activity levels in people with chronic pain. Describe and explore the characteristics and relationships of these participants in terms of pain severity, fear of movement, patterns of activity, anxiety and depression, and number and differing types of long term conditions and how these all correlate with PA levels. Explore PA levels of chronic pain patients and the correlation of psychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with pain lasting more than 12 weeks (chronic pain)
* 16 years or older

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire - Short Form | Entire duration of study- 6 months
  The International Physical Activity Questionnaire -Short Form measures free-living physical activity levels. The questionnaire is psychometrically tested and used as an instrument to measure physical activity over the previous seven days of participants. It was developed in 1998 to investigate physical activity levels based on the global standard. The IPAQ short form has demonstrated to have acceptable measurement properties for use in a variety of settings. The nine item instrument asks for time spent in walking, moderate and vigorous intensity physical activity of at least 10-minute durations.

SECONDARY OUTCOMES:
Demographics questionnaire | Entire duration of study - 6 months
  The demographics questionnaire will collect information about the participants' age, gender, nationality, ethnicity, duration of condition, living environment.
Brief Pain Inventory - Short Form | Entire duration of study - 6 months
  The Brief Pain Inventory - Short Form (BPI-SF) is a widely used questionnaire used with persons with chronic non-malignant painful conditions. It is composed of a nine-item self-administered questionnaire to evaluate the severity of an individuals' pain and impact on their daily function. The BPI-SF required participants to rate their current pain intensity, pain in the last 24 hours at its worst, least and average by using a numerical scale of 0-10. Participants are also asked to rate the extent to which their pain interferes with seven quality of life domains. The scales to these domains are bound by words "does not interfere" and "interferes completely". The reliability has been reported in several chronic pain conditions.
The Patterns of Activity Measure - Pain | Entire duration of study - 6 months
  The Patterns of Activity Measure -Pain (POAM-P) measures pacing/pattern of activity. The questionnaire is composed of 30 self-reported items developed by Cane et al 2007 to measure three activity patterns; avoidance, overdoing and pacing in patients with chronic pain. Each subscale consists of 10 items, where participants are given instructions such as: "People who have pain use different ways to do their daily activity. This about how you do your daily activity". Participants will then rate the statement as to the extent it applies to them on a five-point scale ranging from 0 (not at all) to 4 (always), each subscale ranges in score from 0-40. The POAM-P scale for pacing has shown acceptable psychometric properties.
The Tampa Scale of Kinesiophobia | Entire duration of study - 6 months
  The Tampa Scale of Kinesiophobia (TSK) is a 17 item self-completed questionnaire that will be used to assess the subjective rating of kinesiophobia or fear of movement. The TSK was originally developed to differentiate between non-excessive fear and phobia among patients with musculoskeletal pain. It has been deemed a valid and reliable psychometric measure used for pain relating to different body parts. The scores of the questionnaire ranged from 17 to 68 where higher scores indicate a higher degree of kinesiophobia.
The Depression, Anxiety and Stress Scale - 42 | Entire duration of study - 6 months
  The Depression, Anxiety and Stress Scale - 42 (DASS-42) is a 42-item self-report instrument that consists of three scales that assess three negative emotional states of depression, anxiety and stress over the last week. Each of the 42 items has four responses ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). The DASS42 requires participants to respond to statements immediately in relation to their feelings of the previous week. Higher scores relate to higher levels of depression, anxiety or stress. Previous findings showed that DASS42 has reliable psychometric properties in relation to internal consistency, convergent and discriminant validity in clinical and non-clinical populations.

CONTACTS AND LOCATIONS:
Overall Officials: Chee Wee Tan, PhD, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No